CLINICAL TRIAL: NCT05801302
Title: Acute Effects of Different Foam Rolling Protocols on the Plantar Flexors' Musculotendinous Properties in Healthy Individuals
Brief Title: Effects of Foam Rolling on the Plantar Flexors' Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Jeam Marcel Geremia, Dr, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 4436122
Record Dates: First submitted 2023-03-10; First posted 2023-04-06 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Foam Roller; Achilles Tendon

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Raters and outcomes assessor will be blinded to the participants' allocation in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foam rolling (longer volume) (Experimental): Participants will perform a single session with a longer foam rolling volume. The protocol will be 3 sets of 60 seconds, with between-sets intervals of 30 seconds and a standardized command to the participant to perform the highest pressure possible. The speed will be controlled through metronome (30 bpm). The foam rolling will be performed with the foam roller placed under the plantar flexors and Achilles tendon in a sitting position, with hands supported to the ground, keeping the body out of contact with the ground, with the unassessed leg crossed above the leg of interest. A standard device (smooth foam roller) with dimensions of 30 cm x 15 cm will be used.
  Interventions: Device: Foam rolling (longer volume)
- Foam rolling (shorter volume) (Active Comparator): Participants will perform a single session with a shorter foam rolling volume. The protocol will be 3 sets of 30 seconds, with between-sets intervals of 30 seconds and a standardized command to the participant to perform the highest pressure possible. The speed will be controlled through metronome (30 bpm). The foam rolling will be performed with the foam roller placed under the plantar flexors and Achilles tendon in a sitting position, with hands supported to the ground, keeping the body out of contact with the ground, with the unassessed leg crossed above the leg of interest. A standard device (smooth foam roller) with dimensions of 30 cm x 15 cm will be used.
  Interventions: Device: Foam rolling (shorter volume)
- Control condition (No Intervention): Participants will remain in the intervention position (in a sitting position, with hands supported to the ground, with the unassessed leg crossed above the leg of interest) for 180 seconds (longer volume time), without the application of any intervention

INTERVENTIONS:
Device: Foam rolling (shorter volume) — A single intervention will be performed (3 sets of 30 seconds, with between-sets intervals of 30 seconds).
  Arms: Foam rolling (shorter volume)
Device: Foam rolling (longer volume) — A single intervention will be performed (3 sets of 60 seconds, with between-sets intervals of 30 seconds).
  Arms: Foam rolling (longer volume)

SUMMARY:
Self-massage is a set of therapeutic techniques performed by the individual using instruments such as a foam roller (i.e., foam rolling [FR]). This technique has been used in rehabilitation to recover myofascial dysfunctions and in physical/sports training, to improve performance in functional and sports activities. Possible changes in the muscle's and tendon's mechanical properties may help to explain the FR effects, however, the dose-response relationship is not clear acutely. Furthermore, body composition also seems to influence the pressure applied to the different tissues during FR, since it can attenuate the forces applied on the tissues. Therefore, the aim of this study is to verify the acute effects of different FR volumes on the plantar flexors' musculotendinous properties in healthy individuals. Twenty healthy subjects (male and female) aged between 18-35 years will perform three different FR conditions: FR90 (3x30s), FR180 (3x60s), and a control condition (CTRL; without the application of any intervention) with a seven-day wash-out period. The Achilles tendon morphological, mechanical, and material properties, medial gastrocnemius passive muscular stiffness, plantar flexors' muscle architecture, and the adipose tissue's thickness, skin temperature and the jump height (assessed during the unilateral countermovement jump) will be obtained. Assessments will be carried out before and immediately after the FR application in the different conditions. Descriptive statistics (mean, standard deviation, and standard error) will be used to present the results. The normality and sphericity of the data will be evaluated using the Shapiro-Wilk and Mauchly tests, respectively. A two-way ANOVA (condition [FR90, FR180, and CTRL] and moments [pre- and post-intervention]) will be used to compare the results. A post-hoc Bonferroni test will be used to find possible differences. A Pearson product-moment correlation test (parametric data) or a Spearman correlation test (non-parametric data) will be used to verify the association between the adipose tissue's thickness and the evaluated parameters. The effect size (Cohen's d) of each condition will be obtained. Responsiveness to conditions (FR90, FR180, and CTRL) will be determined using the typical error.

DETAILED DESCRIPTION:
Self-massage is a set of therapeutic technique performed by the individual using instruments such as a foam roller (i.e., foam rolling [FR]). This technique has been used in rehabilitation to recover myofascial dysfunctions and in physical/sports training, to improve performance in functional and sports activities. Possible changes in the muscle's and tendon's mechanical properties may help to explain the FR effects. Although some studies have found a decreased muscle stiffness after FR intervention, other studies have reported no changes in muscle stiffness. Furthermore, a single study investigated the FR effects on the tendon and found no stiffness changes post-intervention. The between-studies methodological procedures heterogeneity, especially the different FR protocols (e.g., pressure-volume) may partially justify conflicting results. However, the dose-response relationship is not clear acutely. Furthermore, body composition also seems to influence the pressure applied to the different tissues during FR. Therefore, the aim of this study is to verify the acute effects of different FR volumes on the plantar flexors' musculotendinous properties in healthy individuals. Twenty healthy subjects (male and female) aged between 18-35 years will perform three different FR conditions: FR90 (3x30s), FR180 (3x60s), and a control condition (CTRL; without the application of any intervention) with a seven-day wash-out period. The weight-bearing during the FR application will be obtained through ground reaction forces, measured through force platform. The Achilles tendon morphological properties (length and cross-sectional area) will be evaluated using ultrasonography. In order to evaluate the mechanical (stiffness, force, and elongation) and material (Young's modulus, stress, and strain) properties, three maximum voluntary isometric contractions (MVIC) will be performed in a plantar flexion ramp in the isokinetic dynamometer with ultrasonography. The tendon force will be corrected by the tibialis anterior coactivation and adjusted by the tendon displacement caused by joint rotation during MVIC. The tendon elongation will be monitored during CMVIC using the ultrasound. The medial gastrocnemius muscle stiffness will be calculated by the variation in a passive dorsiflexion torque (isokinetic dynamometer) and the variation in the muscle length (ultrasound). The adipose tissue's thickness also will be obtained from ultrasound. The skin temperature will be evaluated by a thermographic camera to investigate possible post-intervention changes. The unilateral countermovement jump performance will be evaluated by 2D kinematic data measurements, using a video camera. Assessments will be carried out before and immediately after the FR application in the different conditions. Descriptive statistics (mean, standard deviation, and standard error) will be used to present the results. The normality and sphericity of the data will be evaluated using the Shapiro-Wilk and Mauchly tests, respectively. A two-way ANOVA (condition [FR90, FR180, and CTRL] and moments [pre- and post-intervention]) will be used to compare the results. A post-hoc Bonferroni test will be used to localize possible differences. A Pearson product-moment correlation test (parametric data) or a Spearman correlation test (non-parametric data) will be used to verify the association between the adipose tissue's thickness on the evaluated parameters, classified as none (0.0), weak (0.1-0.3), moderate (0.4-0.6), strong (0.7-0.9), or perfect (1.0). The effect size (Cohen's d) of each condition will be obtained, classified as small effect size (< 0.20); moderate effect size (0.20-0.50); or large effect size (>0.80). Responsiveness to conditions (FR90, FR180, and CTRL) will be determined using the typical error.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female;
* Age between 18 and 35 years;
* Not involved in strength training for lower limbs;
* Not using foam rolling regularly;
* Only women using hormonal contraceptive pills will be included in order to standardize the hormonal cycle.

Exclusion Criteria:

* History in the last year of musculoskeletal injuries in the lower limbs that represent a contraindication for the execution of maximum exercises or that may interfere with performance during evaluations and treatment sessions (Achilles tendinopathy, ligament ruptures with or without surgical procedures, recent cases of muscle injury or sprain of ankle);
* Presenting with inflammation, acute pain or delayed muscle pain on the day of assessment;
* Performing some type of high-intensity physical activity for up to 72 hours before assessments;
* Ingestion of some type of analgesic medication, alcohol or caffeine in the last 48 hours before the evaluations;
* Have respiratory or cardiovascular conditions considered a risk factor or limiting to maximum tests;
* Use of anabolic steroid supplements.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Changes in Achilles tendon stiffness | Change from baseline at immediately after intervention
  Tendon stiffness will be obtained by calculating the slope in the last 10% of the linear region of the force-deformation curve.
Changes in medial gastrocnemius passive muscular stiffness | Change from baseline at immediately after intervention
  The medial gastrocnemius stiffness will be calculated by the variation in passive torque (dorsiflexion) divided by the variation in muscle length (assessed by ultrasound).
Changes in unilateral countermovement jump height | Change from baseline at immediately after intervention
  The unilateral countermovement jump height will be measured using video camera and Tracker software.

SECONDARY OUTCOMES:
Changes in tendon Young's modulus | Change from baseline at immediately after intervention
  Tendon elastic modulus (Young's modulus) will be obtained by calculating the slope in the last 10% of the linear region of the stress-strain curve.
Changes in Achilles tendon cross-sectional area | Change from baseline at immediately after intervention
  To obtain the Achilles tendon cross-sectional area (CSA), the ultrasound probe will be placed perpendicular to the tendon (in the transverse plane), and 3 images will be obtained with reference to the distances of 2, 4, 6, 8 and 10 cm of the muscle insertion in the calcaneus bone. Area values will be obtained for each image, and the final value of the area will be calculated by the average of these five values.
Changes in Achilles tendon length | Change from baseline at immediately after intervention
  To obtain Achilles tendon length, the ultrasound probe will be placed longitudinally to the tendon (in the sagittal plane). The most distal portion of the Achilles tendon, inserted into the calcaneus bone, will be determined by ultrasound, and the respective point will be marked on the skin. After this, the probe will be moved to a proximal position until the visualization of the medial gastrocnemius myotendinous junction (MTJ), which is also marked on the skin. The distance between the two marked points on the skin will be measured with a measuring tape, this distance being considered representative of the tendon length.
Changes in muscle Architecture | Change from baseline at immediately after intervention
  Muscular architecture will be evaluated with an ultrasound. Muscle architecture parameters will involve fascicle length, pennation angle, muscle thickness, and the adipose tissue's thickness. The images will be obtained with the subjects in the ventral decubitus position on a stretcher, with the knees extended and the ankle in neutral position (heel line at a 90° angle with respect to the longitudinal axis of the leg, 0° of plantarflexion). A custom system will be used to secure the ankle in the neutral position. The probe will be positioned longitudinally to the muscle fibers at 30% proximal for medial and lateral gastrocnemius, and 50% for soleus, of the distance between the popliteal fold and the lateral malleolus center.
Changes in skin temperature | Change from baseline at immediately after intervention
  The skin temperature (plantar flexors and Achilles tendon region) will be evaluated using a thermographic camera.

CONTACTS AND LOCATIONS:
Overall Officials: Jeam Geremia, Dr, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided